CLINICAL TRIAL: NCT02026765
Title: Clinical Outcomes About Heparin Surface Modified Aspheric Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Dr, Wenzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5AT-6M
Record Dates: First submitted 2013-12-17; First posted 2014-01-03 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Inflammatory Reaction
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin Surface Modified Aspheric Lens (Other): Heparin Surface Modified Aspheric Lens
  Interventions: Device: heparin surface modified aspheric lens
- traditional lens (Other): traditional Aspheric lens
  Interventions: Device: traditional lens

INTERVENTIONS:
Device: traditional lens — A random eyes with traditional lens
  Arms: traditional lens
Device: heparin surface modified aspheric lens — the other eye implant heparin surface modified aspheric lens
  Arms: Heparin Surface Modified Aspheric Lens

SUMMARY:
The purpose of this study is to obverse the effect of this type lens in the same as traditional aspheric intraocular lens at the same time, whether can further improve the effects of operation.

DETAILED DESCRIPTION:
1. Heparin surface treatment lens can reduce inflammatory reaction.
2. Modified aspheric lens are more in line with human optical properties than the traditional aspheric lens.
3. To obverse the effect of this type lens in the same as traditional aspheric intraocular lens at the same time, whether can further improve the effects of operation.
4. After one day, one week, one month, three month follow-up，Key observation on the flare, the optical quality, contrast sensitivity and other parameters.Study the postoperative inflammatory reaction with test group lens，and the impact on the visual quality.

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients

Exclusion Criteria:

* Eyed patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
flare value in the anterior chamber after surgery | six months
  use Laser Flare Meter to measure the flare in the anterior chamber to evaluate postoperative ocular inflammatory reaction

SECONDARY OUTCOMES:
the ocular and the anterior corneal aberration after surgery | six months
  use wavefront aberrometer to measure the ocular and the anterior corneal aberration to evaluate postoperative ocular optical quality

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD. PhD., Study Director — Wenzhou Medical University
Locations (1):
- The Affiliated Eye hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China